CLINICAL TRIAL: NCT07245290
Title: Effect of Local Infiltration of Liposomal Bupivacaine on Postoperative Analgesia in Patients With Craniotomy Microvascular Decompression: a Randomized Controlled Study
Brief Title: Effect of Local Infiltration of Liposomal Bupivacaine on Postoperative Analgesia in Patients With Craniotomy Microvascular Decompression
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-1230
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Liposomal Bupivacaine; Microvascular Decompression
Keywords: Liposomal Bupivacaine; Microvascular decompression; scalp infiltration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): For this group of patients, after routine disinfection and draping, the incision operation was performed directly.
  Interventions: Other: normal operation
- Liposome bupivacaine group (Experimental): After the patients in this group underwent preoperative disinfection and draping, the surgical doctor gradually infiltrated the liposomal bupivacaine into the incision layer by layer (subcutaneous → muscle → periosteum), and then proceeded with the incision operation.
  Interventions: Drug: liposomal bupivacaine local infiltration

INTERVENTIONS:
Drug: liposomal bupivacaine local infiltration — Before the operation, local infiltration of the scalp incision was performed using liposomal bupivacaine.
  Arms: Liposome bupivacaine group
Other: normal operation — Following the normal procedure, after direct disinfection and draping, the incision operation can be carried out.
  Arms: Control group

SUMMARY:
Background: Approximately 60-84% of patients undergoing craniotomy experience moderate to severe pain within 48 hours postoperatively, with posterior fossa craniotomy patients experiencing more severe pain. Microvascular decompression (MVD) is a type of posterior fossa surgery. Traditional analgesic regimens rely on intravenous opioids, but these have significant side effects. Currently, local infiltration at the incision site is a simple and effective analgesic method in multimodal analgesia protocols after craniotomy. Liposomal bupivacaine (Exparel®) is a new type of sustained-release local anesthetic. Its liposome encapsulation technology can extend the drug release time to 72 hours, covering the entire time window of postoperative acute pain and helping patients better control pain.

Objective: This study aims to explore the efficacy of local infiltration of liposomal bupivacaine at the scalp incision in acute pain after microvascular decompression in neurosurgery and provide evidence for clinical practice.

Methods: This study is a single-center, prospective, randomized controlled trial. A total of 100 patients scheduled for elective craniotomy for microvascular decompression will be enrolled. They will be randomly assigned to the liposomal bupivacaine incision infiltration group (LB group) or the conventional treatment control group (C group). After induction of general anesthesia, in the LB group, after preoperative disinfection and draping, the surgeon will perform layer-by-layer infiltration of the incision (subcutaneous → muscle → periosteum) before skin incision. In the C group, the routine procedure of direct disinfection and draping followed by skin incision will be performed. Both groups will receive standardized multimodal analgesia after returning to the ward. The primary outcome measure is the area under the curve of the numerical rating scale (NRS) for rest pain from 0 to 72 hours postoperatively (AUC NRS-R0-72). Secondary outcome measures include the time to first analgesic request within 72 hours postoperatively; rescue analgesia within 72 hours postoperatively (opioid analgesics converted to morphine milligram equivalents); NRS scores at 6, 12, 24, 48, and 72 hours postoperatively; hemodynamic data: heart rate and blood pressure at skin incision, 1 hour after skin incision, 2 hours after skin incision, at the end of surgery, and 1 hour postoperatively; QoR-15 score at 72 hours postoperatively; and length of hospital stay and hospitalization costs.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years old;
* (2) ASA classification ≤ III grade, patients scheduled to undergo craniotomy and microvascular decompression surgery.

Exclusion Criteria:

* (1) Trauma or emergency patients;
* (2) Patients with cardiac conduction block (sinus node conduction block or atrioventricular conduction block);
* (3) Patients with coagulation dysfunction;
* (4) Patients who have abused alcohol or had severe dependence on anesthetic drugs within the past 2 months;
* (5) Patients with uncontrolled anxiety disorder, schizophrenia or other mental illnesses;
* (6) Patients with a history of allergy to local anesthetics or non-steroidal drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
AUC NRS-R0-72 | From 0 to 72 hours after the operation
  The area under the curve of the resting pain score from 0 to 72 hours after the operation

SECONDARY OUTCOMES:
The time required for the first postoperative analgesic administration within 72 hours after the operation | From 0 to 72 hours after the operation
  The time required for the first postoperative analgesic administration within 72 hours after the operation
The situation of emergency pain relief within 72 hours after the operation | From 0 to72 hours after the operation
  The situation of emergency pain relief within 72 hours after the operation(Converting the dosage of opioid painkillers into milligram equivalents of morphine)
NRS scores at 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours after the operation | From 0 to 72 hours after the operation
  Numerical rating scale（NRS) scores at 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours after the operation
Hemodynamic data 1 | From the time of incision to 1 hour after surgery
  Heart rate at the time of incision, 1 hour after incision, 2 hours after incision, at the end of the surgery, and 1 hour after surgery.
Hemodynamic data 2 | From the time of incision to 1 hour after surgery
  Blood pressure at the time of incision, 1 hour after incision, 2 hours after incision, at the end of the surgery, and 1 hour after surgery.
QoR-15 score | At 72 hours after the operation
  The 15-item quality of recovery scale at 72 hours after the operation
Length of hospital stay | From admission to discharge
  The duration from admission to discharge
Hospital expenses | From admission to discharge
  The medical expenses incurred from admission to discharge

IPD SHARING:
Plan to Share IPD: No